CLINICAL TRIAL: NCT03372590
Title: NEO Rehabilitation Program for Premature Infants at Risk for Cerebral Palsy
Brief Title: NEO Rehab for Infants at Risk of Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Santina Zanelli, Associate Professor of Pediatrics, University of Virginia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20318
Record Dates: First submitted 2017-12-08; First posted 2017-12-13 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Prematurity; Cerebral Palsy
Keywords: general movement assessment
MeSH Terms: conditions — Premature Birth; Cerebral Palsy | interventions — Kangaroo-Mother Care Method; Massage; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NICU-based rehabilitation bundle (Experimental): Patients identified to be at high risk for cerebral palsy will be enrolled after parental consent is obtained to the NICU rehabilitation program. This program consists of maternal-driven evidence based intervention that include: vocal soothing, scent exchange, comforting touch, kangaroo care, and infant massage. These intervention will be provided at GA-appropriate intervals.
  Interventions: Other: NICU-based rehabilitation bundle
- Standard of care (Other): Infants not participating in the intervention study will be provided with standard or care. Interventions include kangaroo care, physical therapy and infant massage provided by NICU staff.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: NICU-based rehabilitation bundle — Maternal-driven gestational age-appropriate intervention/activity bundle, including the evidence-based elements of vocal soothing, comforting touch, scent exchange, kangaroo care, and infant massage
  Other Names: scent exchange; kangaroo care; massage; vocal soothing; comforting touch
  Arms: NICU-based rehabilitation bundle
Other: Standard of care — Standard NICU care
  Arms: Standard of care

SUMMARY:
Premature infants are at increased risk of developing cerebral palsy (CP). Early interventions for at risk infants have the potential to decrease disease severity and improve quality of life. All infants demonstrate general movements (GMs), which are reliable indicators of brain function and can be reproducibly evaluated using the General Movement Assessment (GMA) tool.

Prior studies have demonstrated the impact of early maternal-driven intervention strategies on neurodevelopmental outcomes in preterm infants. Investigators have shown that interventions promoting the establishment of emotional connection between the infant and his or her mother, including mother/infant calming sessions with scent cloth exchange, vocal soothing, eye contact, and kangaroo care, can impact neurodevelopmental outcomes at 18 months. Investigators have also shown that 60 minutes of kangaroo care leads to decreasing levels of the stress hormone cortisol in both mothers and infants.

This pilot study aims to determine the feasibility of a maternal-driven early intervention bundle in preterm infants with abnormal GMA.

DETAILED DESCRIPTION:
The study objective are 3-fold:

1. To determine the proportion of infants (<32 weeks gestation and/or <1500g) who have abnormal GMs findings using the GMA tool.
2. To determine the feasibility of NICU based rehabilitation program in 20 infants determined to be at high risk for CP using the GMA tool. The intervention bundle will consist of a maternal-driven gestational age (GA)-appropriate intervention bundle that will include evidence-based interventions including vocal soothing, comforting touch, scent exchange, kangaroo care, and infant massage. Patients will be compared to contemporary and GA-matched controls receiving standard of care with a 1:2 assignment.
3. To evaluate the short-term impact of a maternal-driven intervention bundle on the mother-infant dyad. Maternal stress will be measured using the Parental Stress Scale for NICU patients (PSS: NICU) prior to the intervention and prior to the infant's NICU discharge. Further, stress will be assessed by measuring maternal and infant salivary cortisol pre-and post-kangaroo care on 3 separate occasions (post enrollment in the study, mid-hospital stay, and prior to discharge). Measures of maternal anxiety and depression will be evaluated prior to the intervention and prior to NICU discharge using the Patient Reported Outcomes Measurement Information System (PROMIS) instrument.

The investigators hypothesize that the intervention will lead to positive and measurable outcomes for the mother-infant dyad.

ELIGIBILITY:
Inclusion Criteria:

* Infant Gestational age <32 weeks AND/OR birth weight <1500g

Exclusion Criteria:

* Any clinical condition / diagnosis that would restrict the ability of the mother to do Kangaroo Care per the current UVA Kangaroo Care guideline
* Non-English-speaking mother
* Mother is a prisoner
* Confirmed inability to return for follow-up appointment

Max Age: 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2018-09-02 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
NICU-based rehabilitation program feasibility | 2 years
  The feasibility of a maternal driven intervention bundle will be assessed using a maternal diary and unannounced observations. The ability to perform the required intervention greater than 75% of the time will be considered successful

SECONDARY OUTCOMES:
Evolution of GMA patterns in high risk infants | 2 years
  GME will be scored on enrollment and at NICU discharge
Impact on maternal stress and depression | 2 years
  Assessed on enrollment and NICU discharge using the PSS-NICU and PROMIS instrument

CONTACTS AND LOCATIONS:
Overall Officials: Santina A Zanelli, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided